CLINICAL TRIAL: NCT03439904
Title: Impact of Individualized Pharmaceutical-care on Medication Adherence and Outcome of Cancer Pain in Opioid-tolerant Outpatients
Brief Title: Individualized Pharmaceutical-care in Outpatients With Cancer Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Ping Huang, Chief of Pharmacy, Zhejiang Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ECCOPG-003
Record Dates: First submitted 2018-02-14; First posted 2018-02-20 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Cancer Pain
Keywords: pharmaceutical care; adherence
MeSH Terms: conditions — Cancer Pain | interventions — Pharmaceutical Services

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pharmaceutical care intervention group (Experimental): Patients will receive individualized pharmaceutical care in addition to usual medical care
  Interventions: Other: Pharmaceutical care
- control group (No Intervention): Patients will receive usual medical care

INTERVENTIONS:
Other: Pharmaceutical care — Patients receive pharmaceutical care including individualized evaluation and intervention of adherence, efficacy and safety in cancer pain treatment.
  Arms: pharmaceutical care intervention group

SUMMARY:
The purpose of the study is to investigate the impact of pharmaceutical care on cancer pain treatment for opioid-tolerant outpatients

DETAILED DESCRIPTION:
This study is a prospective multicenter randomized controlled study to investigate the impact of pharmaceutical care on cancer pain treatment for opioid-tolerant outpatients treated with sustained released morphine, oxycodone, and transdermal fentanyl.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older;
* Histologically confirmed solid tumor;
* Diagnosed chronic cancer pain;
* Opioid-tolerant patients;
* Overall survival is expected to be over 3 months;
* Karnofsky performance score≥50;
* Willing and able to comply with the protocol

Exclusion Criteria:

* Patients aged 18 years or older;
* Histologically confirmed solid tumor;
* Diagnosed chronic cancer pain;
* Opioid-tolerant patients;
* Overall survival is expected to be over 3 months;
* Karnofsky performance score≥50;
* Willing and able to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-06-30 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in medication adherence | Change from baseline at 1 month
  The investigators will measure the change in medication adherence via Morisky Scale from baseline to 1 months. Morisky Scale contains 4 questions, and the total score ranges from 0 to 4 with lower scores indicating higher adherence.

SECONDARY OUTCOMES:
Change in pain score | Change from baseline pain score at 1 month
  Comparison of pain score of cancer pain patients with or without pharmaceutical care. Pain score will be assessed using numeric rating scale (NRS). An NRS allows a person to describe the intensity of his/her pain as a number usually ranging from 0 to 10, where "0" means "no pain" and "10" means pain as "bad as it could be."
Change in quality of life | Change from baseline quality of life at 1 month
  Comparison of quality of life of cancer pain patients with or without pharmaceutical care. Quality of life is assessed using EuroQol- 5 Dimension (EQ-5D). It is a questionnaire to measure quality of life. It contains 5 domains: Mobility; Self-care; Usual activity; Pain; Anxiety/depression. It also contains a visual analogue scale. Weights are used to score the responses to the 5 domains, with scores ranging from 0 to 1 (where a score of 1 represents a perfect state). For the visual analogue scale, participants draw a line from a box to the point on the thermometer-like scale corresponding to their health state, 0-100 (100 = Best health state)
Change in patients' knowledge of cancer pain and analgesics | Change from baseline knowledge at 1 month
  Comparison of knowledge of cancer pain and analgesics for cancer pain patients with or without pharmaceutical care. Knowledge of pain treatment and analgesics will be assessed using investigator designed questionnaire. This questionnaire consists of 16 items assessing patients' knowledge about cancer pain, treatment of cancer pain and medications for cancer pain. The total score ranges from 0 to 16 with higher score indicating better knowledge.
Incidence of adverse events [safety and tolerability] | Up to 1 month
  Adverse events will be assessed throughout the study according the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Event (CTCAE) Version 4.0. Number and percentage of subjects who experienced an adverse event in this study is presented.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Ding H, Song Y, Wu N, Zheng X, Wei Q, Sun Y, Xie R, Zhai Q, Xu S, Qi Y, Wang Y, Li H, Yang L, Fan Q, Zhao Q, Chen J, Shi J, Duan C, Du Q, Zhang Y, Song Z, Fu S, Cai Y, Huang X, Fang L, Liu Y, Huang P. Impact of individualized pharmaceutical care on efficacy and safety of opioid-tolerant outpatients with cancer pain: a multicenter randomized controlled trial. Ann Transl Med. 2022 Sep;10(18):989. doi: 10.21037/atm-22-4091. PMID 36267757